CLINICAL TRIAL: NCT02627573
Title: Randomized Trial of GVHD Prophylasxis With Post-transplantation Cyclophocphomide (PTCy) or Thymoglobulin in Unrelated SCT Recepients With Chronic Myeloproliferative Neoplasms and Myelodisplatic Syndrome
Brief Title: Trial of GVHD Prophylasxis With PTCy or Thymoglobulin in Unrelated SCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Head of adolescent and adult department of oncology, heamatology and transplantation, St. Petersburg State Pavlov Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06/15-n
Record Dates: First submitted 2015-12-04; First posted 2015-12-11 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Leukemia, Chronic Myeloid; Myelodysplastic Syndromes; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative
Keywords: Cyclophosphamide; Thymoglobulin; Myelodysplastic Syndromes; Immunosuppressive Agents; Immune System Diseases; Busulfan; Fludarabine; Tacrolimus; Mycophenolate mofetil; Antineoplastic Agents, Alkylating; Myeloablative Agonists; Hematopoietic Stem Cell Transplantation; Allogeneic Transplantation; Leukemia, Chronic Myeloid; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Immune System Diseases | interventions — Busulfan; fludarabine phosphate; Tacrolimus; Mycophenolic Acid; Cyclophosphamide; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thymoglobulin (Experimental): Days -7 through -2: Fludarabine 30 mg/m2/day iv x 6 days Days -6 through -5 Busulfan 1 mg/kg po qid x 2 days Days -4 through -3 Thymoglobulin 2,5 mg/kg po qd x 2 days Days -1 through +30: Mycophenolate mofetil 30 mg/kg/day, maximum 2 g/day, iv or po x 30 days Days -1 through +150: Tacrolimus 0.03 mg/kg/day with further correction by concentration
  Interventions: Procedure: Unrelated allogeneic stem cell transplantation; Drug: Busulfan; Drug: Fludarabine monophosphate; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Thymoglobulin
- PTCy (Experimental): Days -7 through -2: Fludarabine 30 mg/m2/day iv x 6 days Days -4 through -3: Busulfan 1 mg/kg po qid x 2 days Day 0: Infusion of unmanipulated graft Day +3 and +4: Cyclophosphamide 50 mg/kg/day iv Days +5 through +35: Mycophenolate mofetil 30 mg/kg/day, maximum 2 g/day, iv or po x 30 days Days +5 through +120: Tacrolimus 0.03 mg/kg/day with further correction by concentration
  Interventions: Procedure: Unrelated allogeneic stem cell transplantation; Drug: Busulfan; Drug: Fludarabine monophosphate; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: Cyclophosphamide

INTERVENTIONS:
Procedure: Unrelated allogeneic stem cell transplantation
Drug: Busulfan
Drug: Fludarabine monophosphate
Drug: Tacrolimus
Drug: Mycophenolate mofetil
Drug: Cyclophosphamide
  Arms: PTCy
Drug: Thymoglobulin
  Arms: Thymoglobulin

SUMMARY:
Purpose There is a growing evidence of high efficacy of post-transplantation cyclophocphomide (PTCy)-based GVHD prophylaxis in haploidentical and matched related and unrelated bone marrow transplantation. There is limitted, but growing data on safety and efficacy of this prophylaxis in unrelated and peripheral blood stem cell transplantations. Use of PTCy in chronic myeloproliferative neoplasms and myelodisplatic syndrome is of particular interest. On the one hand, PTCy could reduce the incidence of chronic GVHD and long-term bormidity. On the other hand, there is a concern, that PTCy can increase the incidence of graft failures in this group of patients. Currently published data indicate that low-dose Thymoglobulin-based prophylaxis is the most promissing compatitor in terms of acute and chronic GVHD control. So there is a rationale to randomize Thymoglobulin and PTCy as GVHD prophilaxis. Pre-transplant assesment of moratlity (PAM)-index will be used as the strata for randomization, as it is the paramter that takes into account the most important factors effecting survival. The conditioning regimen and the other two components of GVHD prophylaxis (mycophenolate mofetil and tacrolimus) will be identical in the two arms of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an indication for allogeneic hematopoietic stem cell transplantation
* Diagnosis: Chronic myeloid leukemia Myelodysplastic Syndromes Myeloprolipherative neoplsm unclassified Atypical chronic myelogenous leukemia
* Signed informed consent
* Patients with 10/10 HLA-matched unrelated donor available. The donor and recipient must be identical by the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1. Mismatches in these loci are not allowed.
* Peripheral blood stem cells as graft source
* No second tumors
* No prior history of Thymoglobulin exposure or no history of anaphylactic shock after Thymoglobulin administration
* No severe concurrent illness

Exclusion Criteria:

* Moderate or severe cardiac dysfunction, left ventricular ejection fraction <50%
* Moderate or severe decrease in pulmonary function, FEV1 <70% or DLCO<70% of predicted
* Respiratory distress >grade I
* Severe organ dysfunction: AST or ALT >5 upper normal limits, bilirubin >1.5 upper normal limits, creatinine >2 upper normal limits
* Creatinine clearance < 60 mL/min
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Incidence of primary graft failure | 60 days

SECONDARY OUTCOMES:
Incidence of acute GVHD, grades II-IV | 365 days
Incidence of chronic GVHD, moderate and severe (NIH criteria) | 365 days
Non-relapse mortality analysis | 365 days
Event-free survival analysis | 365 days
Overall survival analysis | 365 days
Relapse rate analysis | 365 days
Toxicity (NCI CTCAE 4.03) | 100 days
  Toxicity parameters based on NCI CTCAE 4.03 grades: hepatotoxicity (liver function tests), nephrotoxicity (creatinine), neurotoxicity (attending physician assessment), mucositis (attending physician assessment), hemorrhagic cystitis (attending physician assessment), cardiotoxicity (ECG, echocardiography). Additional toxicity parameters: incidence and severity of veno-occlusive disease, incidence of transplant-associated microangiopathy
Infectious complications, including analysis of severe bacterial, fungal and viral infections incidence | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Boris V. Afanasyev, Professor, Principal Investigator — First Pavlov State Medical University of St. Petersburg
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No